CLINICAL TRIAL: NCT03715465
Title: The Clinical Utility of DLMO in the Treatment of Delayed Sleep-Wake Phase Disorder: A Randomized Trial
Brief Title: The Clinical Utility of Measuring the Circadian Clock in Treatment of Delayed Sleep-Wake Phase Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: American Academy of Sleep Medicine (Other)
Responsible Party: Principal Investigator, Leslie Swanson, Clinical Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00145052
Record Dates: First submitted 2018-10-19; First posted 2018-10-23 (Actual); Results first posted 2022-11-25 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-10

CONDITIONS: Delayed Sleep Phase Syndrome
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Estimated DLMO (Active Comparator): Four weeks (28 days) of nightly melatonin 0.5 mg fast dissolve tablets timed to be administered 3 hours before estimated dim light melatonin onset.
  Interventions: Drug: Melatonin 0.5 MG
- Measured DLMO (Experimental): Four weeks (28 days) of nightly melatonin 0.5 mg fast dissolve tablets timed to be administered 3 hours before measured dim light melatonin onset.
  Interventions: Drug: Melatonin 0.5 MG; Other: Dim Light Melatonin Onset (salivary)

INTERVENTIONS:
Drug: Melatonin 0.5 MG — Melatonin tablet
Other: Dim Light Melatonin Onset (salivary) — Test to determine the time of melatonin onset in saliva under dim light conditions
  Arms: Measured DLMO

SUMMARY:
This study will test whether measuring the circadian clock during treatment of delayed sleep-wake phase disorder results in greater improvements in sleep compared to estimating the circadian clock.

DETAILED DESCRIPTION:
The study is a randomized, controlled, parallel double-blind 4-week trial of 0.5 mgs of exogenous melatonin timed to either 3 h before actual dim light melatonin onset (DLMO) based on in-home measurement (M-DLMO, n = 25) or 3 h before DLMO estimated at 2 h before average sleep onset time based on actigraphy and sleep diary (E-DLMO, n = 25) in adult participants with delayed sleep-wake phase disorder. All participants will receive melatonin 0.5 mgs. Outcomes include change in DLMO, subjective and objective sleep parameters, and daytime symptoms.

As of January 7, 2020, the Insomnia Severity Index was removed from the IRB-approved protocol. No data were collected for this measure.

ELIGIBILITY:
Inclusion Criteria:

* Meet diagnostic criteria for delayed sleep wake phase disorder
* Female participants of childbearing potential must agree to use a reliable method of contraception from the screening visit until 4 weeks after the study has completed.

Exclusion Criteria:

* Hypersensitivity to melatonin or any other component of the product
* Sleep disorder other than delayed sleep wake phase disorder
* Medical and psychiatric conditions that may influence sleep or be affected by melatonin
* Current use of medications which may have interactions with melatonin
* Pregnancy or breastfeeding
* Routine night shift work
* Past month travel or planned travel during the study across more than one time zone
* Use of melatonin in the past month
* Current use of medications that may interfere with the measurement of melatonin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2021-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Swanson, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Swanson LM, de Sibour T, DuBuc K, Conroy DA, Raglan GB, Lorang K, Zollars J, Hershner S, Arnedt JT, Burgess HJ. Low-dose exogenous melatonin plus evening dim light and time in bed scheduling advances circadian phase irrespective of measured or estimated dim light melatonin onset time: preliminary findings. J Clin Sleep Med. 2024 Jul 1;20(7):1131-1140. doi: 10.5664/jcsm.11076. PMID 38445651

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 44 participants total were enrolled in this trial, 4 of whom withdrew before randomization to the arms.
Period: Overall Study
Arm/Group | Measured DLMO | Estimated DLMO
Started | 20 | 20
Completed | 19 | 18
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Measured DLMO | Estimated DLMO | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.45 (6.19) | 26.70 (5.62) | 26.08 (5.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 29
  Male | 4 | 7 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 11 | 18 | 29
  Black/African American | 4 | 0 | 4
  Asian | 4 | 0 | 4
  I have two or more racial backgrounds | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 19 | 19 | 38
  Hispanic or Latino | 0 | 1 | 1
  Ethnicity Unknown | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 40
Dim Light Melatonin Onset [Mean (Standard Deviation); unit: Clock time in hours] — Onset of melatonin in dim light conditions as measured in saliva (also called DLMO). Time of DLMO is measured in clock time. Population: Baseline DLMO was not calculable for 5 participants in the E-DLMO group
  Clock time in hours
    number analyzed (Participants) | 20 | 15 | 35
    (all) | 22.90 (2.23) | 22.55 (1.52) | 22.75 (1.93)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Time of Dim Light Melatonin Onset (DLMO) at 4 Weeks
Description: Onset of melatonin in dim light conditions as measured in saliva (also called DLMO). Time of DLMO is measured in clock time and change in time of DLMO is measured in hours. The change score is calculated as time at 4 weeks minus baseline time. Thus, positive scores indicate a shift towards a later onset of melatonin and negative scores indicate a shift towards an earlier onset of melatonin.
Time Frame: After 4 weeks of melatonin therapy
Population: Data were not analyzed for 2 participants in the Measured DLMO group and 7 participants in the Estimated DLMO group due to missing or incalculable DLMO data at one or both of the time points.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Measured DLMO | Estimated DLMO
Number analyzed (Participants) | 18 | 13
Hours | -1.23 (1.53) | -1.58 (1.30)
Statistical Analysis 1: Comparison: Measured DLMO vs Estimated DLMO; Test type: Superiority; p = 0.510, t-test, 2 sided

2. Secondary Outcome: Change From Baseline Score on Wrist Actigraphy and Self-Report Diary Sleep Diary Parameters - Total Sleep Time at 4 Weeks
Description: Change in total sleep time is measured in hours. The change score is calculated by subtracting total sleep time at 4 weeks from total sleep time at baseline. Thus, positive scores indicate an increase in total sleep time, whereas negative scores indicate a decrease in total sleep time.
Time Frame: After 4 weeks of melatonin therapy
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Measured DLMO | Estimated DLMO
Number analyzed (Participants) | 19 | 18
Hours
  change in total sleep time per diary | 0.41 (0.79) | 0.65 (0.99)
  change in total sleep time per actigraphy | 0.63 (0.79) | 0.66 (1.00)
Statistical Analysis 1: Comparison: Measured DLMO vs Estimated DLMO; Per diary; Test type: Superiority; p = 0.411, t-test, 2 sided
Statistical Analysis 2: Comparison: Measured DLMO vs Estimated DLMO; Per wrist actigraphy; Test type: Superiority; p = 0.920, t-test, 2 sided

3. Secondary Outcome: Change From Baseline Score on Wrist Actigraphy and Self-Report Diary Sleep Diary Parameters - Sleep Onset Time at 4 Weeks
Description: Sleep onset time is measured in clock time and reflects time of falling asleep. The change score is calculated as time at 4 weeks minus baseline time. Thus, positive scores indicate a shift towards a later fall asleep time and negative scores indicate a shift towards an earlier fall asleep time.
Time Frame: After 4 weeks of melatonin therapy
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Measured DLMO | Estimated DLMO
Number analyzed (Participants) | 19 | 18
Hours
  change in sleep onset time per diary | -1.73 (1.10) | -1.84 (1.40)
  change in sleep onset time per actigraphy | -1.58 (1.11) | -1.63 (1.47)
Statistical Analysis 1: Comparison: Measured DLMO vs Estimated DLMO; Per diary; Test type: Superiority; p = 0.787, t-test, 2 sided
Statistical Analysis 2: Comparison: Measured DLMO vs Estimated DLMO; Per wrist actigraphy; Test type: Superiority; p = 0.916, t-test, 2 sided

4. Secondary Outcome: Change From Baseline Score on Wrist Actigraphy and Self-Report Diary Sleep Diary Parameters - Sleep Offset Time at 4 Weeks
Description: Sleep offset time is measured in clock time and reflects time of waking for the day. The change score is calculated as time at 4 weeks minus baseline time. Thus, positive scores indicate a shift towards a later wake time and negative scores indicate a shift towards an earlier wake time.
Time Frame: After 4 weeks of melatonin therapy
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Measured DLMO | Estimated DLMO
Number analyzed (Participants) | 19 | 18
Hours
  change in sleep offset time per diary | -1.61 (0.98) | -1.96 (0.96)
  change in sleep offset time per actigraphy | -1.15 (0.89) | -1.45 (1.18)
Statistical Analysis 1: Comparison: Measured DLMO vs Estimated DLMO; Per diary; Test type: Superiority; p = 0.270, t-test, 2 sided
Statistical Analysis 2: Comparison: Measured DLMO vs Estimated DLMO; Per wrist actigraphy; Test type: Superiority; p = 0.406, t-test, 2 sided

5. Secondary Outcome: Change From Baseline Score on Wrist Actigraphy and Self-Report Diary Sleep Onset Latency at 4 Weeks
Description: Length of time to sleep onset latency in minutes (reflects time to fall asleep). The change score is calculated as time at 4 weeks minus baseline time. Thus, a negative scores indicate a reduction in time to fall asleep, whereas positive scores indicate an increase in time to fall asleep.
Time Frame: After 4 weeks of melatonin therapy
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Measured DLMO | Estimated DLMO
Number analyzed (Participants) | 19 | 18
Minutes
  change in sleep onset latency per diary | -14.35 (32.61) | -10.21 (17.25)
  change in sleep onset latency per actigraphy | -9.75 (36.83) | -0.53 (25.19)
Statistical Analysis 1: Comparison: Measured DLMO vs Estimated DLMO; Per diary; Test type: Superiority; p = 0.635, t-test, 2 sided
Statistical Analysis 2: Comparison: Measured DLMO vs Estimated DLMO; Per wrist actigraphy; Test type: Superiority; p = 0.383, t-test, 2 sided

6. Secondary Outcome: Change From Baseline Score on Epworth Sleepiness Scale at 4 Weeks
Description: Self-report of daytime sleepiness. Scores range from 0 to 24. Scores of 10 or higher indicate excessive daytime sleepiness. The change score is calculated as score at 4 weeks minus baseline score.Thus, positive scores indicate an increase in sleepiness, whereas negative scores indicate a reduction in sleepiness.
Time Frame: After 4 weeks of melatonin therapy
Population: One participant in the Measured DLMO group was not included in the analysis because they did not complete the measure at one of the time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Measured DLMO | Estimated DLMO
Number analyzed (Participants) | 18 | 18
score on a scale | -1.61 (2.75) | -0.78 (3.80)
Statistical Analysis 1: Comparison: Measured DLMO vs Estimated DLMO; Test type: Superiority; p = 0.456, t-test, 2 sided

7. Secondary Outcome: Change From Baseline Score on Multidimensional Fatigue Inventory at 4 Weeks
Description: Self-report of daytime fatigue. Scores range from 20-100; higher scores indicate more fatigue. The change score is calculated as score at 4 weeks minus baseline score. Thus, positive scores indicate an increase in fatigue, whereas negative scores indicate a reduction in fatigue.
Time Frame: After 4 weeks of melatonin therapy
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Measured DLMO | Estimated DLMO
Number analyzed (Participants) | 18 | 18
score on a scale | -3.78 (8.73) | -6.50 (10.43)
Statistical Analysis 1: Comparison: Measured DLMO vs Estimated DLMO; Test type: Superiority; p = 0.402, t-test, 2 sided

8. Secondary Outcome: Change From Baseline Score on Sheehan Disability Scale at 4 Weeks
Description: Self-report of functional impairment in works/school, social, and family life. Scores range from 0-30; higher scores indicate more impairment.
  The change score is calculated as time at 4 weeks minus baseline time Thus, positive scores indicate increased impairment, whereas negative scores indicate a reduction in impairment.
Time Frame: After 4 weeks of melatonin therapy
Population: 10 participants in the Measured DLMO and 5 participants in the Estimated DLMO group did not complete this measure due to an error in data collection procedures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Measured DLMO | Estimated DLMO
Number analyzed (Participants) | 9 | 13
score on a scale | -0.33 (4.92) | -5.85 (6.63)
Statistical Analysis 1: Comparison: Measured DLMO vs Estimated DLMO; Test type: Superiority; p = 0.047, t-test, 2 sided

9. Secondary Outcome: Change From Baseline Score on Patient Health Questionnaire-9 at 4 Weeks
Description: Self-report of depression symptoms. Scores range from 0-27; higher scores indicate more severe depression. The change score is calculated as score at 4 weeks minus baseline score. Thus, positive scores indicate an increase in depression, whereas negative scores indicate a reduction in depression.
Time Frame: After 4 weeks of melatonin therapy
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a Questionnaire
Arm/Group | Measured DLMO | Estimated DLMO
Number analyzed (Participants) | 18 | 18
Score on a Questionnaire | 0.28 (2.63) | -0.39 (3.53)
Statistical Analysis 1: Comparison: Measured DLMO vs Estimated DLMO; Test type: Superiority; p = 0.525, t-test, 2 sided

10. Secondary Outcome: Change From Baseline Score on Generalized Anxiety Disorder-7 Scale at 4 Weeks
Description: Self-report of generalized anxiety symptoms. Scores range from 0-21; higher scores indicate more severe anxiety. The change score is calculated as score at 4 weeks minus baseline score. Thus, positive scores indicate an increase in anxiety, whereas negative scores indicate a reduction in anxiety.
Time Frame: After 4 weeks of melatonin therapy
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Measured DLMO | Estimated DLMO
Number analyzed (Participants) | 18 | 18
units on a scale | 1.11 (3.03) | -0.50 (2.79)
Statistical Analysis 1: Comparison: Measured DLMO vs Estimated DLMO; Test type: Superiority; p = 0.106, t-test, 2 sided

11. Secondary Outcome: Change From Baseline Score on the Pittsburgh Sleep Quality Index at 4 Weeks
Description: Self-report of sleep quality. Seven subscale scores are summed to obtain a global score. Global scores range from 0 to 21; scores of 5 or higher indicate poor sleep quality. The change score is calculated as score at 4 weeks minus baseline score. Thus, positive scores indicate a worsening of sleep quality, whereas negative scores indicate an improvement in sleep quality.
Time Frame: After 4 weeks of melatonin therapy
Population: One participant in the Measured DLMO and one participant in the Estimated DLMO group were not included in the analysis because they did not complete the measure at one of the time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Measured DLMO | Estimated DLMO
Number analyzed (Participants) | 18 | 17
score on a scale | 1.61 (2.87) | -0.59 (3.74)
Statistical Analysis 1: Comparison: Measured DLMO vs Estimated DLMO; Test type: Superiority; p = 0.059, t-test, 2 sided

12. Secondary Outcome: Change From Baseline Score on the Morningness Eveningness Questionnaire at 4 Weeks
Description: Self-report of chronotype. Scores range from 16-86. Lower scores indicate more eveningness.The change score is calculated as score at 4 weeks minus baseline score. Thus, positive scores indicate a shift towards more morningness, whereas negative scores indicate a shift towards more eveningness.
Time Frame: After 4 weeks of melatonin therapy
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Measured DLMO | Estimated DLMO
Number analyzed (Participants) | 18 | 18
score on a scale | 4.89 (4.73) | 12.17 (9.65)
Statistical Analysis 1: Comparison: Measured DLMO vs Estimated DLMO; Test type: Superiority; p = 0.007, t-test, 2 sided

13. Secondary Outcome: Change From Baseline Score on the PROMIS-Sleep Disturbance Scale at 4 Weeks
Description: Self-report of sleep disturbances. Scores range from 8-40. Higher scores indicate greater sleep disturbance. The change score is calculated as score at 4 weeks minus baseline score. Thus, positive scores indicate a worsening of sleep disturbance, whereas negative scores indicate an improvement in sleep disturbance.
Time Frame: After 4 weeks of melatonin therapy
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Measured DLMO | Estimated DLMO
Number analyzed (Participants) | 18 | 18
score on a scale | -3.56 (6.28) | -5.94 (5.85)
Statistical Analysis 1: Comparison: Measured DLMO vs Estimated DLMO; Test type: Superiority; p = 0.246, t-test, 2 sided

14. Secondary Outcome: Change From Baseline Score on the PROMIS-Sleep Related Impairment Scale at 4 Weeks
Description: Self-report of impairment related to sleep. Scores range from 8-40. Higher scores indicate greater impairment due to sleep.
  The change score is calculated as score at 4 weeks minus baseline score. Thus, positive scores indicate an increase in impairment due to sleep, whereas negative scores indicate a reduction in impairment due to sleep.
Time Frame: After 4 weeks of melatonin therapy
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Measured DLMO | Estimated DLMO
Number analyzed (Participants) | 18 | 18
score on a scale | -3.94 (5.25) | -6.11 (7.75)
Statistical Analysis 1: Comparison: Measured DLMO vs Estimated DLMO; Test type: Superiority; p = 0.333, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 4 weeks.
Arm/Group | Measured DLMO | Estimated DLMO
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 16/20 | 16/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Measured DLMO (N=20) | Estimated DLMO (N=20)
Hypoacusis (Ear and labyrinth disorders) | 0 | 2
Eye irritation (Eye disorders) | 0 | 2
Gingival bleeding (Gastrointestinal disorders) | 0 | 2
Decreased appetite (General disorders) | 2 | 2
Dizziness (Nervous system disorders) | 0 | 2
Headaches (Nervous system disorders) | 4 | 4
Migraine (Nervous system disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 4
Depression (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 3 | 4
Irritability (Psychiatric disorders) | 0 | 2
Somnolence (Psychiatric disorders) | 11 | 9
Rash (Skin and subcutaneous tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-18): https://cdn.clinicaltrials.gov/large-docs/65/NCT03715465/Prot_SAP_000.pdf